CLINICAL TRIAL: NCT02729727
Title: Clinical Study to Evaluate the CryoBalloon™ Full Ablation System for the Ablation of Human Esophageal Epithelium in Patients Undergoing Esophagectomy
Brief Title: Clinical Study to Evaluate CryoBalloon™ Ablation System in Patients Undergoing Esophagectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pentax Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP-0008
Record Dates: First submitted 2016-03-14; First posted 2016-04-06 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2018-01

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Other): To evaluate safety and treatment effect of the CryoBalloon Ablation System for the Ablation of human esophageal epithelium in patients scheduled to undergo esophagectomy
  Interventions: Device: CryoBalloon Ablation System

INTERVENTIONS:
Device: CryoBalloon Ablation System — Tissue Ablation using CryoBalloon Ablation System

SUMMARY:
To evaluate the safety and treatment effect of the CryoBalloon™ Full Ablation System for the ablation of human esophageal epithelium in patients scheduled to undergo esophagectomy

DETAILED DESCRIPTION:
The primary outcomes for the study are the safety and treatment effect of the CryoBalloon™ Ablation System. An esophagectomy will be performed as scheduled following the ablation procedure; histopathological analysis of surgically-resected specimens will be performed to determine the treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* Up to two (2) areas of 3 cm each non-ulcerated, columnar lined esophagus or squamous linted tissue suitable for ablation
* Older than 18 years of age at the time of consent
* Requires a clinically-necessary esophagectomy for esophageal cancer
* Patient has provided written informed consent using the Informed Consent Form approved by the Institution's reviewing Medical Ethics Committee (MEC)

Exclusion Criteria:

* Patient refuses or is unable to provide written informed consent
* Patient has esophageal narrowing limiting access to the intended site of ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06-24 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Safety of CryoBalloon Ablation System | through study completion, an average of 2 weeks
  Incidence of device related serious adverse events

SECONDARY OUTCOMES:
Device Performance | through study completion, an average of 2 weeks
  Ease of deployment of the CryoBalloon, procedure time, endoscope compatibility, device malfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques J.G.H.M. Bergman, MD, PhD, Principal Investigator — AMC Medical Research B.V.
Locations (1):
- Academic Medical Centre Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided